CLINICAL TRIAL: NCT01971541
Title: A Non-inferiority Trial of MBSR and CPT for PTSD
Brief Title: Groups for Regaining Our Wellbeing (GROW)
Acronym: GROW
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 12-112
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: mindfulness; behavior therapies, cognitive; posttraumatic stress disorder; group therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Mindfulness-Based Stress Reduction; 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Stress Reduction (MBSR) (Experimental): An 8-week program designed to teach mindfulness skills
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Cognitive Processing Therapy (Active Comparator): A group-administered PTSD treatment program.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — A validated 8-week group program that teaches mindfulness meditation
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction (MBSR)
Behavioral: Cognitive Processing Therapy — A validated group program of PTSD treatment, which focuses on cognitive processing.
  Other Names: CPT
  Arms: Cognitive Processing Therapy

SUMMARY:
The proposed study is a randomized, controlled trial that will assess whether two group interventions for PTSD - Mindfulness-Based Stress Reduction (MBSR) and Cognitive Processing Therapy-Cognitive only (CPT-C) result in similar improvements in PTSD symptoms and health-related quality of life (QOL). One hundred fifty-two Veterans with PTSD will be randomized to MBSR (n = 76) or CPT-C (n = 76). Comprehensive assessments will take place post-treatment and 3 months later.

DETAILED DESCRIPTION:
The proposed study is a randomized, controlled non-inferiority trial that will assess whether Mindfulness-Based Stress Reduction (MBSR) and Cognitive Processing Therapy-Cognitive only (CPT-C) result in equivalent improvement in both PTSD symptoms and health-related quality of life (QOL). PTSD symptoms will be measured by the Clinician Administered PTSD Scale - CAPS and health-related QOL will be measured by the SF-36V Mental Component Summary Score - MCS. In an exploratory aim, we will also assess whether there is a clinically meaningful response as defined by improvement in both PTSD symptoms and QOL (defined as a reliable change of 12 points on the CAPS and 10 points on the MCS, respectively, according to the reliable change index).7, 8 One hundred fifty-two Veterans with PTSD will be randomized to MBSR (n = 76) or CPT-C (n = 76). Comprehensive assessments will take place post-treatment and 3 months later. Qualitative analysis of brief semi-structured interview data will be used to identify previously unrecognized factors pertaining to participation, adherence and response to treatment, spirituality and religion as treatment moderators, and to identify common themes that may inform treatment retention efforts for both MBSR and CPT-C. In addition, potential moderators of change in PTSD symptoms and QOL for MBSR and CPT-C will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with current DSM-V diagnosis of PTSD

Exclusion Criteria:

* Current substance use disorder other than alcohol,
* Alcohol involvement that poses a safety concern or is associated with inability to follow through on assessments and class attendance as evinced by past month appointment attendance record in CPRS,
* Suicidal or homicidal ideation with intent or plan within the past 3 months,
* Self harm in the past 3 months,
* A psychotic disorder,
* Uncontrolled bipolar disorder,
* Chart diagnoses of borderline personality disorder or antisocial personality disorder,
* In-patient admission for psychiatric reasons within the past month,
* Prior participation in MBSR or CPT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
PTSD symptoms | 3 months follow-up
  Clinician-administered PTSD Scale (CAPS)

SECONDARY OUTCOMES:
Health-related Quality of Life | 3 months follow-up
  SF-36V

CONTACTS AND LOCATIONS:
Overall Officials: David J. Kearney, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States